CLINICAL TRIAL: NCT05414019
Title: Evaluation of Root Resorption Following Different Mandibular Incisors Intrusive Mechanics : A Randomized Clinical Trial
Brief Title: Evaluation of Root Resorption Following Different Mandibular Incisors Intrusive Mechanics
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud Salah Mahmoud Ali Nassar, Principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 799/2234
Record Dates: First submitted 2022-05-29; First posted 2022-06-10 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Orthodontic Tooth Movement; Intrusion of Tooth; Resorption, Root
Keywords: Intrusion; Root resorption; Cone beam computed tomography; Utility Arch; Nitinol reverse curve wire; Miniscrew; Mandibular incisors
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Intervention Model Description: The total sample of patients will be randomly divided into three equal groups: Miniscrew: 7 patients will receive an intrusive force delivered by elastics from 2 miniscrews between mandibular lateral incisor and mandibular canine. Utility arch: 7 patients will receive an intrusive force delivered by intrusive utility arch. Nitinol reverse curve wire: 7 patients will receive an intrusive force delivered by Nitinol reverse curve wire.
Masking Description: Observation:
  Each patient will be followed up on periodic base for progress evaluation and integrity checks, as well as root resorption will be evaluated using CBCT images taken before and after the intrusion.
  Ethical considerations:
  An informed consent form (attached copy) that explains every step in the research will be given and discussed carefully with the patient and his/her parents before participation in the study and should be signed freely. The objectives of the study will be discussed and explained with the patients and / or their guardians and they will receive a copy of the consent form as well.
  Data management and analysis:
  The data will be collected, tabulated, and statistically analyzed using Statistical Package for Social Sciences (SPSS program, version 18, Inc., Chicago, III).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mini-screw (Active Comparator): 7 patients will receive an intrusive force delivered by elastics from 2 mini-screws between mandibular lateral incisor and mandibular canine.
  Interventions: Other: Mini-screw
- Utility arch (Active Comparator): 7 patients will receive an intrusive force delivered by intrusive utility arch.
  Interventions: Other: Utility arch
- Nitinol reverse curve wire (Active Comparator): 7 patients will receive an intrusive force delivered by Nitinol reverse curve wire.
  Interventions: Other: Nitinol reverse curve wire

INTERVENTIONS:
Other: Mini-screw — 7 patients will receive an intrusive force delivered by elastics from 2 mini-screws between mandibular lateral incisor and mandibular canine.
  Arms: Mini-screw
Other: Utility arch — 7 patients will receive an intrusive force delivered by intrusive utility arch.
  Arms: Utility arch
Other: Nitinol reverse curve wire — 7 patients will receive an intrusive force delivered by Nitinol reverse curve wire
  Arms: Nitinol reverse curve wire

SUMMARY:
Evaluation of root resorption following different mandibular incisors intrusive mechanics : A randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patient will be included in this study if has:

  * An age range between 12 and 16 years.
  * Deep overbite with excessive curve of Spee of more than 5mm
  * Over erupted lower incisors.
  * Permanent teeth are all present (except for third molar).
  * No previous orthodontic treatment.
  * No indications or symptoms of periodontal disease in the past or present, as determined by clinical and radiographic examination

Exclusion Criteria:

* Patients who needed surgery to fix skeletal problems.
* Any previous trauma or root canal therapy
* Missing lower incisor.
* Patients with congenital dentoskeletal disorders

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Linear amount of root resorption | Change in Linear Root resorption at 6 months
  Cone beam computed tomography linear measurements
Volumetric amount of root resorption | Change in Volumetric Root resorption at 6 months
  Cone beam computed tomography volumetric measurements

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Nassar, student, Principal Investigator — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Egypt

REFERENCES:
- [Background] Goel P, Tandon R, Agrawal KK. A comparative study of different intrusion methods and their effect on maxillary incisors. J Oral Biol Craniofac Res. 2014 Sep-Dec;4(3):186-91. doi: 10.1016/j.jobcr.2014.11.007. Epub 2014 Dec 6. PMID 25737942
- [Background] Hamdan AM, Lewis SM, Kelleher KE, Elhady SN, Lindauer SJ. Does overbite reduction affect smile esthetics? Angle Orthod. 2019 Nov;89(6):847-854. doi: 10.2319/030819-177.1. Epub 2019 Jul 15. PMID 31306077
- [Background] Piancino MG, Tortarolo A, Di Benedetto L, Crincoli V, Falla D. Chewing Patterns and Muscular Activation in Deep Bite Malocclusion. J Clin Med. 2022 Mar 19;11(6):1702. doi: 10.3390/jcm11061702. PMID 35330027
- [Background] Nielsen IL. Vertical malocclusions: etiology, development, diagnosis and some aspects of treatment. Angle Orthod. 1991 Winter;61(4):247-60. doi: 10.1043/0003-3219(1991)0612.0.CO;2. PMID 1763835
- [Background] Sonnesen L, Svensson P. Temporomandibular disorders and psychological status in adult patients with a deep bite. Eur J Orthod. 2008 Dec;30(6):621-9. doi: 10.1093/ejo/cjn044. Epub 2008 Aug 5. PMID 18684706
- [Background] Guven BA, Ciger S. Evaluation of the Effect of Fixed Anterior Biteplane Treatment on Temporomandibular Joint in Patients with Deep Bite. Turk J Orthod. 2020 Mar 1;33(1):8-12. doi: 10.5152/TurkJOrthod.2020.19108. eCollection 2020 Mar. PMID 32284893
- [Background] Millett DT, Cunningham SJ, O'Brien KD, Benson PE, de Oliveira CM. Orthodontic treatment for deep bite and retroclined upper front teeth in children. Cochrane Database Syst Rev. 2018 Feb 1;2(2):CD005972. doi: 10.1002/14651858.CD005972.pub4. PMID 29390172
- [Background] Nanda R. The differential diagnosis and treatment of excessive overbite. Dent Clin North Am. 1981 Jan;25(1):69-84. No abstract available. PMID 6937401
- [Background] Burstone CR. Deep overbite correction by intrusion. Am J Orthod. 1977 Jul;72(1):1-22. doi: 10.1016/0002-9416(77)90121-x. PMID 267433